CLINICAL TRIAL: NCT03588429
Title: The Ratio of Hypnotic to Analgesic Potency of Volatile Anesthetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018CZTCWM
Record Dates: First submitted 2018-07-06; First posted 2018-07-17 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2018-08

CONDITIONS: Anesthesia
Keywords: Sevoflurane; Isoflurane
MeSH Terms: interventions — Sevoflurane; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sevoflurane (Experimental): Anesthesia was maintained with sevoflurane.
  Interventions: Drug: Sevoflurane
- Isoflurane (Experimental): Anesthesia was maintained with isoflurane.
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Sevoflurane — Anesthesia was maintained with sevoflurane in patients undergoing standardized nociceptive stimulus (long-lasting tetanic stimulus of the ulnar nerve; 30 s, 50 mA, 50 Hz, square-wave).
  Other Names: SEVO
  Arms: Sevoflurane
Drug: Isoflurane — Anesthesia was maintained with isoflurane in patients undergoing standardized nociceptive stimulus (long-lasting tetanic stimulus of the ulnar nerve; 30 s, 50 mA, 50 Hz, square-wave).
  Other Names: ISO
  Arms: Isoflurane

SUMMARY:
The aim of this clinical trial is to evaluate the ratio of hypnotic to analgesic potency of sevoflurane and isoflurane at equi-minimum alveolar concentration using EEG analysis.

DETAILED DESCRIPTION:
Anesthetic agents vary in their relative hypnotic potency. Recent studies demonstrated that equi-minimum alveolar concentration of various volatile anesthetic agents may produce different spectral entropy or bispectral index values. However, there is no study that demonstrate the difference between analgesic potency of volatile anesthetics. The aim of this clinical trial is to evaluate the ratio of hypnotic to analgesic potency of sevoflurane and isoflurane at equi-minimum alveolar concentration using EEG analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing general anesthesia using volatile anesthetics and intubation
* patients with american society of anesthesiologist physical status I, II
* patients obtaining written informed consent

Exclusion Criteria:

* patients with a history of any psychiatric or neurological disease
* patients who had received any medication affecting the central nervous system
* patients who had received medication affecting the sympathetic or parasympathetic nervous systems
* patients undergoing supraglottic airway for airway management
* pregnant women

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
qCON index | the 10 min at steady-state anesthesia after endotracheal intubation
  The hypnotic potency of volatile anesthetics was evaluated by qCON index during standardized nociceptive stimulus (30 s, 50 mA, 50 Hz tetanic stimulation).

SECONDARY OUTCOMES:
qNOX index | the 10 min at steady-state anesthesia after endotracheal intubation
  The analgesic potency of volatile anesthetics was evaluated by qNOX index during standardized nociceptive stimulus (30 s, 50 mA, 50 Hz tetanic stimulation).

CONTACTS AND LOCATIONS:
Overall Officials: Ruizhao Lv, M.D, Principal Investigator — Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine
Locations (1):
- Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine, Cangzhou, Hebei, China